CLINICAL TRIAL: NCT01488890
Title: Evaluation of the Immune Response to Different Schedules of a Tetravalent Dengue Vaccine Administered With or Without Yellow Fever Vaccine in US Adults.
Brief Title: Immune Response to Different Schedules of a Tetravalent Dengue Vaccine Given With or Without Yellow Fever Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYD51; U1111-1122-1892 (Other: WHO)
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Fever; Dengue Hemorrhagic Fever; Yellow Fever
Keywords: Dengue fever; Dengue Hemorrhagic Fever; CYD dengue vaccine; Yellow Fever; Flavivirus
MeSH Terms: conditions — Dengue; Severe Dengue; Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CYD Dengue vaccine: Group 1 (Experimental): Participants received 3 doses of CYD dengue vaccine; one each at 0, 6 and 12 months.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus
- CYD Dengue vaccine: Group 2 (Experimental): Participants received 3 doses of CYD dengue vaccine; one each at 0, 2 and 6 months.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus
- CYD Dengue and Yellow Fever vaccine: Group 3 (Experimental): Participants received 3 doses of CYD dengue vaccine; one each at 0, 2 and 6 months, and single dose of YF vaccine at Day 0.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus; Biological: Yellow Fever
- Yellow Fever vaccine: Group 4 (Active Comparator): Participants received single dose of YF vaccine at Day 0.
  Interventions: Biological: Yellow Fever

INTERVENTIONS:
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus — 0.5 mL, Subcutaneous
  Other Names: CYD Dengue Vaccine
  Arms: CYD Dengue vaccine: Group 1
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus — 0.5 mL, Subcutaneous
  Other Names: CYD Dengue Vaccine
  Arms: CYD Dengue vaccine: Group 2
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus — 0.5 mL, Subcutaneous
  Other Names: CYD Dengue Vaccine
  Arms: CYD Dengue and Yellow Fever vaccine: Group 3
Biological: Yellow Fever — 0.5 mL, Subcutaneous
  Other Names: YF VAX®
  Arms: CYD Dengue and Yellow Fever vaccine: Group 3; Yellow Fever vaccine: Group 4

SUMMARY:
The aim of this study was to evaluate the administration of CYD dengue vaccine serotypes (1, 2, 3 and 4) following a compressed schedule in 3 different populations.

Primary Objectives:

* To describe the humoral immune response to each of the 4 parental dengue virus serotypes at baseline and 28 days after CYD dengue vaccine Dose 3 in Group 1 (Month [M] 13) and Group 2 (M07), irrespective of whether or not Yellow Fever (YF) vaccine has been previously administered.
* To describe the persistence of the humoral immune response to each of the 4 parental dengue virus serotypes 6 months after CYD dengue vaccine Dose 3 in Group 1 (M18) and Group 2 (M12), irrespective of whether or not YF vaccine has been previously administered.

Secondary Objective:

* To describe the humoral immune response to each of the 4 parental dengue virus serotypes at baseline and 28 days after CYD dengue vaccine Dose 1 and Dose 2 in Groups 1 and 2, irrespective of whether or not YF vaccine has been previously administered.
* To describe the humoral immune response to each of the 4 parental dengue virus serotypes at baseline and 28 days after CYD dengue Dose 1 in the combined YF-participants in Group 1 (N=60) and Group 2 (N=60), and in Group 3 (N=120).
* To describe by FV status at baseline the humoral immune response to each of the 4 parental dengue virus serotypes at baseline and 28 days after each injection of CYD dengue vaccine in Groups 1, 2, and 3.
* To describe the safety profile after each injection of CYD dengue vaccine and/or YF vaccine.

DETAILED DESCRIPTION:
Participants were randomized to 4 different groups to receive either CYD dengue vaccine and/or YF vaccine. Participants who already received YF vaccine prior to enrolment were randomized to one of the 2 groups receiving CYD dengue vaccine alone. Participants were evaluated for immunogenicity, antibody persistence, reactogenicity and safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 18 to <= 45 years on the day of inclusion
* Informed consent form had been signed and dated
* Able to attend all scheduled visits and complied with all trial procedures
* For participants classified as YF positive (+) to be included in Groups 1 and 2, previous vaccination (3 months to 10 years) with YF vaccine confirmed by acceptable documentation.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination)
* Participation in the 4 weeks preceding the first trial vaccination, or planned participation during the present trial period, in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks following each trial vaccination
* For all participants classified as YF negative (-), any previous vaccination against Flavivirus (FV) diseases (including Japanese Encephalitis [JE], tick-borne encephalitis, and YF)
* For participants classified as YF+, previous vaccination against FV diseases except YF (including JE and tick-borne encephalitis)
* For all participants, any FV vaccination planned during the trial period outside the study protocol
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Self-reported history of FV infection (e.g., JE, Dengue, YF, West Nile), confirmed either clinically or serologically
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances, including dry natural latex
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Identified as an employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employee or the Investigator
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0°C [>=100.4°F]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Previous residence (> 12 months) in, or travel in the last 30 days to FV endemic regions
* History of thymic pathology (thymoma), thymectomy, or myasthenia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2011-12-06 (Actual); Primary Completion 2013-09-27 (Actual); Study Completion 2013-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (7):
- United States (7):
  - Alabaster, Alabama
  - Sacramento, California
  - Jacksonville, Florida
  - Silver Spring, Maryland
  - Springfield, Missouri
  - Las Vegas, Nevada
  - West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kirstein J, Douglas W, Thakur M, Boaz M, Papa T, Skipetrova A, Plennevaux E. Immunogenicity of the CYD tetravalent dengue vaccine using an accelerated schedule: randomised phase II study in US adults. BMC Infect Dis. 2018 Sep 21;18(1):475. doi: 10.1186/s12879-018-3389-x. PMID 30241510
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 06 December 2011 to 22 March 2012 in the United States.
Pre-assignment Details: A total of 390 participants were enrolled and randomized in the study.
Groups:
- CYD Dengue and Yellow Fever (YF) Vaccine: Group 3: Participants received 3 doses of CYD dengue vaccine; one each at 0, 2 and 6 months, and single dose of YF vaccine at Day 0.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever (YF) Vaccine: Group 3 | Yellow Fever Vaccine: Group 4
Started | 120 | 120 | 120 | 30
Treated | 120 | 120 | 119 | 30
Completed | 88 | 100 | 85 | 25
Not Completed | 32 | 20 | 35 | 5
Not completed — Serious adverse event | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 4 | 0
Not completed — Lost to Follow-up | 13 | 10 | 20 | 3
Not completed — Withdrawal by Subject | 14 | 10 | 11 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3 | Yellow Fever Vaccine: Group 4 | Total
Number analyzed (Participants) | 120 | 120 | 120 | 30 | 390
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 120 | 120 | 30 | 390
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.6 (7.63) | 32.6 (7.32) | 32.6 (7.52) | 34.8 (8.63) | 32.5 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 61 | 60 | 17 | 195
  Male | 63 | 59 | 60 | 13 | 195

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Each Dengue Virus Serotype Following Injection (Inj.) With CYD Dengue Vaccine Dose 3: Group 1 and Group 2
Description: GMTs of antibodies against each dengue virus serotype (parental strain) was assessed using the dengue plaque reduction neutralization test (PRNT).
Time Frame: Pre-injection 1, 28 days and 6 months post-injection 3
Population: Full Analysis Set included participants who received at least 1 Inj. of CYD dengue or/ YF vaccine, had at least 1 blood sample drawn and valid post-Inj. serology result. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected, analyzed for Group 3 and 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2
Number analyzed (Participants) | 117 | 119
Titers (1/dilution)
  Dengue Virus Serotype 1: Pre-injection 1 | 5.38 [4.85 to 5.96] | 5.13 [4.98 to 5.28]
  Dengue Virus Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 93 | 108
  Dengue Virus Serotype 1: 28 days Post-injection 3 | 14.8 [11.3 to 19.4] | 15.9 [12.6 to 20.0]
  Dengue Virus Serotype 1: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 1: 6 months Post-injection 3 | 13.3 [10.2 to 17.4] | 9.01 [7.54 to 10.8]
  Dengue Virus Serotype 2: Pre-injection 1 | 5.19 [4.82 to 5.58] | 5.22 [4.96 to 5.50]
  Dengue Virus Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 94 | 108
  Dengue Virus Serotype 2: 28 days Post-injection 3 | 51.2 [38.2 to 68.6] | 59.9 [45.8 to 78.4]
  Dengue Virus Serotype 2: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 2: 6 months Post-injection 3 | 45.6 [31.6 to 65.6] | 38.7 [29.5 to 50.8]
  Dengue Virus Serotype 3: Pre-injection | 5.32 [4.94 to 5.73] | 5.28 [5.03 to 5.55]
  Dengue Virus Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 94 | 107
  Dengue Virus Serotype 3: 28 days Post-injection 3 | 45.7 [35.0 to 59.8] | 59.3 [47.0 to 74.7]
  Dengue Virus Serotype 3: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 3: 6 months Post-injection 3 | 30.2 [22.8 to 40.2] | 34.5 [27.5 to 43.3]
  Dengue Virus Serotype 4: Pre-injection 1 | 5.78 [5.16 to 6.48] | 5.11 [4.90 to 5.33]
  Dengue Virus Serotype 4: Post-injection 3: number analyzed (Participants) | 94 | 107
  Dengue Virus Serotype 4: Post-injection 3 | 66.8 [50.9 to 87.8] | 83.1 [61.4 to 112]
  Dengue Virus Serotype 4: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 4: 6 months Post-injection 3 | 74.8 [54.9 to 102] | 41.7 [31.2 to 55.9]

2. Primary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following Injection With CYD Dengue Vaccine Dose 3: Group 1 and Group 2
Description: Seropositivity against each dengue virus serotypes (parental strains) was assessed using the dengue PRNT. Seropositive participants were defined as the participants with neutralizing antibody titer >=10 (1/dilution).
Time Frame: Pre-injection 1, 28 days and 6 months post-injection 3
Population: Analysis was performed on Full Analysis Set. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected, analyzed for Group 3 and 4.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2
Number analyzed (Participants) | 117 | 119
percentage of participants
  Dengue Virus Serotype 1: Pre-injection 1 | 1.7 | 2.5
  Dengue Virus Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 93 | 108
  Dengue Virus Serotype 1: 28 days Post-injection 3 | 52.7 | 56.5
  Dengue Virus Serotype 1: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 1: 6 months Post-injection 3 | 47.7 | 32.7
  Dengue Virus Serotype 2: Pre-injection 1 | 0.9 | 2.5
  Dengue Virus Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 94 | 108
  Dengue Virus Serotype 2: 28 days Post-injection 3 | 84.0 | 88.0
  Dengue Virus Serotype 2: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 2: 6 months Post-injection 3 | 75.0 | 80.8
  Dengue Virus Serotype 3: Pre-injection 1 | 2.6 | 4.2
  Dengue Virus Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 94 | 107
  Dengue Virus Serotype 3: 28 days Post-injection 3 | 85.1 | 90.7
  Dengue Virus Serotype 3: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 3: 6 months Post-injection 3 | 79.5 | 80.8
  Dengue Virus Serotype 4: Pre-injection 1 | 6.8 | 0.8
  Dengue Virus Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 94 | 107
  Dengue Virus Serotype 4: 28 days Post-injection 3 | 88.3 | 86.0
  Dengue Virus Serotype 4: 6 months Post-injection 3: number analyzed (Participants) | 88 | 104
  Dengue Virus Serotype 4: 6 months Post-injection 3 | 86.4 | 74.0

3. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each Dengue Virus Serotype Following Injection With CYD Dengue Vaccine Dose 1 and Dose 2: Group 1 and Group 2
Description: GMTs of antibodies against each dengue virus serotype (parental strain) was assessed using the dengue PRNT.
Time Frame: Pre-injection 1 and 2 and 28 days post-injection 1 and 2
Population: Analysis was performed on Full Analysis Set. Here, 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 3 and 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2
Number analyzed (Participants) | 117 | 119
Titer (1/dilution)
  Dengue Virus Serotype 1: Pre-injection 1 | 5.38 [4.85 to 5.96] | 5.13 [4.98 to 5.28]
  Dengue Virus Serotype 1: 28 days Post-injection 1: number analyzed (Participants) | 117 | 118
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 10.3 [8.15 to 13.1] | 8.75 [7.19 to 10.6]
  Dengue Virus Serotype 1: Pre-injection 2: number analyzed (Participants) | 107 | 118
  Dengue Virus Serotype 1: Pre-injection 2 | 11.2 [8.76 to 14.4] | 11.5 [9.17 to 14.4]
  Dengue Virus Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 101 | 116
  Dengue Virus Serotype 1: 28 days Post-injection 2 | 18.9 [14.3 to 25.1] | 14.9 [11.9 to 18.6]
  Dengue Virus Serotype 2: Pre-injection 1 | 5.19 [4.82 to 5.58] | 5.22 [4.96 to 5.50]
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 30.9 [22.9 to 41.8] | 24.2 [18.0 to 32.4]
  Dengue Virus Serotype 2: Pre-injection 2: number analyzed (Participants) | 106 | 118
  Dengue Virus Serotype 2: Pre-injection 2 | 38.4 [26.2 to 56.1] | 40.0 [28.9 to 55.3]
  Dengue Virus Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 101 | 116
  Dengue Virus Serotype 2: 28 days Post-injection 2 | 64.1 [47.3 to 86.9] | 66.9 [50.9 to 87.9]
  Dengue Virus Serotype 3: Pre-injection 1 | 5.32 [4.94 to 5.73] | 5.28 [5.03 to 5.55]
  Dengue Virus Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 117 | 117
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 32.5 [23.8 to 44.4] | 31.0 [22.9 to 41.8]
  Dengue Virus Serotype 3: Pre-injection 2: number analyzed (Participants) | 107 | 118
  Dengue Virus Serotype 3: Pre-injection 2 | 26.2 [19.3 to 35.5] | 34.5 [25.3 to 47.1]
  Dengue Virus Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 101 | 116
  Dengue Virus Serotype 3: 28 days Post-injection 2 | 47.9 [36.1 to 63.5] | 62.0 [46.8 to 82.2]
  Dengue Virus Serotype 4: Pre-injection 1 | 5.78 [5.16 to 6.48] | 5.11 [4.90 to 5.33]
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 115 | 117
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 121 [74.2 to 197] | 126 [77.5 to 204]
  Dengue Virus Serotype 4: Pre-injection 2: number analyzed (Participants) | 106 | 117
  Dengue Virus Serotype 4: Pre-injection 2 | 60.2 [42.2 to 85.8] | 89.8 [58.6 to 138]
  Dengue Virus Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 101 | 113
  Dengue Virus Serotype 4: 28 days Post-injection 2 | 104 [75.0 to 144] | 111 [78.1 to 159]

4. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following Injection With CYD Dengue Vaccine Dose 1 and Dose 2: Group 1 and Group 2
Description: as for outcome 2
Time Frame: Pre-injection 1 and 2 and 28 days post-injection 1 and 2
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2
Number analyzed (Participants) | 117 | 119
Percentage of participants
  Dengue Virus Serotype 1: Pre-injection 1 | 1.7 | 2.5
  Dengue Virus Serotype 1: 28 days Post-injection 1: number analyzed (Participants) | 117 | 118
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 34.2 | 24.6
  Dengue Virus Serotype 1: Pre-injection 2: number analyzed (Participants) | 107 | 118
  Dengue Virus Serotype 1: Pre-injection 2 | 35.5 | 35.6
  Dengue Virus Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 101 | 116
  Dengue Virus Serotype 1: 28 days Post-injection 2 | 58.4 | 52.6
  Dengue Virus Serotype 2: Pre-injection 1 | 0.9 | 2.5
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 65.0 | 56.3
  Dengue Virus Serotype 2: Pre-injection 2: number analyzed (Participants) | 106 | 118
  Dengue Virus Serotype 2: Pre-injection 2 | 61.3 | 68.6
  Dengue Virus Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 101 | 116
  Dengue Virus Serotype 2: 28 days Post-injection 2 | 86.1 | 87.9
  Dengue Virus Serotype 3: Pre-injection 1 | 2.6 | 4.2
  Dengue Virus Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 117 | 117
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 63.2 | 64.1
  Dengue Virus Serotype 3: Pre-injection 2: number analyzed (Participants) | 107 | 118
  Dengue Virus Serotype 3: Pre-injection 2 | 61.7 | 66.1
  Dengue Virus Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 101 | 116
  Dengue Virus Serotype 3: 28 days Post-injection 2 | 80.2 | 84.5
  Dengue Virus Serotype 4: Pre-injection 1 | 6.8 | 0.8
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 115 | 117
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 67.8 | 67.5
  Dengue Virus Serotype 4: Pre-injection 2: number analyzed (Participants) | 106 | 117
  Dengue Virus Serotype 4: Pre-injection 2 | 71.7 | 67.5
  Dengue Virus Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 101 | 113
  Dengue Virus Serotype 4: 28 days Post-injection 2 | 84.2 | 80.5

5. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each Dengue Virus Serotype Following Injection With CYD Dengue Vaccine Dose 1 In YF Non-Immune Participants: Group 1 and Group 2 (Pooled) and Group 3
Description: GMTs of antibodies against each dengue virus serotype (parental strain) was assessed using the dengue plaque reduction neutralization test-50 (PRNT50). Groups 1 and 2 data was reported as pooled data. YF-non immune participants were defined as participants with YF baseline titer PRNT80 < 10 (1/dilution).
Time Frame: Pre-injection 1 and 28 days post-injection 1
Population: Analysis was performed on Full Analysis Set. Here, "Overall number of participants analyzed = participants evaluable for this outcome measure" and 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected, analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Groups:
- CYD Dengue Vaccine Group 1 and 2: Pooled: All Participants who received 3 doses of CYD dengue vaccine in Group 1 and 2.
Arm/Group | CYD Dengue Vaccine Group 1 and 2: Pooled | CYD Dengue and Yellow Fever Vaccine: Group 3
Number analyzed (Participants) | 116 | 108
Titer (1/dilution)
  Dengue Virus Serotype 1: Pre-injection 1 | 5.19 [4.87 to 5.53] | 5.00 [NA to NA] — The confidence interval (CI) of Geometric Mean was not calculated when standard deviation (SD) = 0.
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 8.71 [7.04 to 10.8] | 7.68 [6.46 to 9.14]
  Dengue Virus Serotype 2: Pre-injection 1 | 5.06 [4.94 to 5.19] | 5.06 [4.94 to 5.20]
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 18.8 [13.9 to 25.3] | 10.8 [8.63 to 13.4]
  Dengue Virus Serotype 3: Pre-injection 1 | 5.21 [4.97 to 5.47] | 5.28 [4.90 to 5.69]
  Dengue Virus Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 114 | 108
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 28.5 [20.4 to 39.7] | 8.88 [7.23 to 10.9]
  Dengue Virus Serotype 4: Pre-injection 1 | 5.43 [4.99 to 5.92] | 5.26 [4.90 to 5.65]
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 114 | 107
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 229 [139 to 378] | 22.6 [15.9 to 32.3]

6. Secondary Outcome: Percentage of YF Non-Immune Participants With Seropositivity Against Each Dengue Virus Serotype Following Injection With CYD Dengue Vaccine Dose 1: Group 1 and Group 2 (Pooled) and Group 3
Description: Seropositivity against each dengue virus serotypes (parental strains) was assessed using the dengue PRNT. Seropositive participants were defined as the participants with neutralizing antibody titer >=10 (1/dilution). Groups 1 and 2 data was reported as pooled data. YF-non immune participants were defined as participants with YF baseline titer dengue plaque reduction neutralization test-80 (PRNT80) <10 (1/dilution).
Time Frame: Pre-injection 1 and 28 days post-injection 1
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Groups:
- CYD Dengue Vaccine Group 1 and Group 2: Pooled: All participants who received 3 doses of CYD dengue vaccine in Group 1 and Group 2.
Arm/Group | CYD Dengue Vaccine Group 1 and Group 2: Pooled | CYD Dengue and Yellow Fever Vaccine: Group 3
Number analyzed (Participants) | 116 | 108
percentage of participants
  Dengue Virus Serotype 1: Pre-injection 1 | 1.7 | 0.0
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 23.3 | 20.4
  Dengue Virus Serotype 2: Pre-injection 1 | 0.9 | 0.9
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 46.6 | 35.2
  Dengue Virus Serotype 3: Pre-injection 1 | 2.6 | 2.8
  Dengue Virus Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 114 | 108
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 57.9 | 25.0
  Dengue Virus Serotype 4: Pre-injection 1 | 3.4 | 1.9
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 114 | 107
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 74.6 | 48.6

7. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each Dengue Virus Serotype Following Each Injection With CYD Dengue Vaccine: Group 1, Group 2 and Group 3 (FV Immune Participants)
Description: GMTs of antibodies against each dengue virus serotype (parental strain) was assessed using the dengue PRNT. FV immune participants were defined as participants with titer >= 10 (1/dilution) for at least 1 serotype with parental dengue virus strain (sera tested by PRNT) or with titer >= 10 (1/dilution) for YF virus (sera with PRNT80 result).
Time Frame: Pre Injection 1, 2 and 3 and 28 days post injection 1, 2 and 3
Population: Analysis was performed on Full Analysis Set. Here, Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3
Number analyzed (Participants) | 63 | 65 | 11
Titer (1/dilution)
  Dengue Virus Serotype 1: Pre-injection 1 | 5.73 [4.72 to 6.94] | 5.23 [4.96 to 5.53] | 14.3 [2.79 to 73.0]
  Dengue Virus Serotype 1: 28 days Post-injection 1: number analyzed (Participants) | 63 | 64 | 11
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 13.9 [9.46 to 20.3] | 9.25 [6.96 to 12.3] | 27.2 [5.96 to 124]
  Dengue Virus Serotype 1: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 1: Pre-injection 2 | 18.0 [11.9 to 27.1] | 12.8 [9.22 to 17.8] | 36.1 [5.89 to 221]
  Dengue Virus Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 53 | 63 | 10
  Dengue Virus Serotype 1: 28 days Post-injection 2 | 25.0 [16.6 to 37.8] | 16.7 [12.6 to 22.2] | 31.4 [8.55 to 115]
  Dengue Virus Serotype 1: Pre-injection 3: number analyzed (Participants) | 51 | 58 | 9
  Dengue Virus Serotype 1: Pre-injection 3 | 12.7 [8.67 to 18.6] | 10.6 [7.98 to 14.1] | 36.3 [5.08 to 260]
  Dengue Virus Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 51 | 59 | 9
  Dengue Virus Serotype 1: 28 days Post-injection 3 | 15.6 [10.6 to 23.0] | 17.2 [12.7 to 23.3] | 79.0 [17.2 to 362]
  Dengue Virus Serotype 2: Pre-injection 1 | 5.35 [4.67 to 6.13] | 5.42 [4.93 to 5.96] | 13.5 [3.71 to 49.4]
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 48.1 [32.8 to 70.5] | 34.4 [23.0 to 51.4] | 66.3 [18.9 to 233]
  Dengue Virus Serotype 2: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 2: Pre-injection 2 | 72.3 [42.3 to 123] | 45.0 [29.8 to 67.9] | 70.2 [18.1 to 272]
  Dengue Virus Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 53 | 63 | 10
  Dengue Virus Serotype 2: 28 days Post-injection 2 | 83.7 [54.6 to 128] | 74.6 [54.5 to 102] | 122 [38.4 to 386]
  Dengue Virus Serotype 2: Pre-injection 3: number analyzed (Participants) | 51 | 60 | 9
  Dengue Virus Serotype 2: Pre-injection 3 | 43.0 [25.9 to 71.3] | 62.3 [42.1 to 92.1] | 63.6 [18.7 to 217]
  Dengue Virus Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 52 | 59 | 9
  Dengue Virus Serotype 2: 28 days Post-injection 3 | 60.0 [39.4 to 91.4] | 68.1 [48.9 to 94.7] | 133 [56.8 to 313]
  Dengue Virus Serotype 3: Pre-injection 1 | 5.61 [4.89 to 6.45] | 5.53 [5.06 to 6.05] | 21.5 [6.05 to 76.2]
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 45.1 [30.5 to 66.8] | 31.2 [21.2 to 46.1] | 98.0 [51.6 to 186]
  Dengue Virus Serotype 3: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 3: Pre-injection 2 | 47.8 [33.0 to 69.2] | 41.1 [27.1 to 62.4] | 105 [27.7 to 396]
  Dengue Virus Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 53 | 63 | 10
  Dengue Virus Serotype 3: 28 days Post-injection 2 | 72.5 [51.6 to 102] | 69.6 [49.9 to 97.0] | 158 [64.1 to 391]
  Dengue Virus Serotype 3: Pre-injection 3: number analyzed (Participants) | 51 | 60 | 9
  Dengue Virus Serotype 3: Pre-injection 3 | 29.9 [20.4 to 43.7] | 48.3 [33.9 to 68.7] | 106 [21.7 to 516]
  Dengue Virus Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 52 | 59 | 9
  Dengue Virus Serotype 3: 28 days Post-injection 3 | 44.8 [31.3 to 64.3] | 71.2 [53.4 to 94.8] | 130 [36.3 to 463]
  Dengue Virus Serotype 4: Pre-injection 1 | 6.55 [5.32 to 8.07] | 5.20 [4.81 to 5.63] | 15.6 [5.33 to 45.6]
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 61 | 65 | 11
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 78.2 [42.4 to 144] | 77.9 [42.1 to 144] | 215 [49.9 to 924]
  Dengue Virus Serotype 4: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 4: Pre-injection 2 | 65.9 [40.8 to 107] | 65.0 [37.9 to 111] | 235 [52.1 to 1059]
  Dengue Virus Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 53 | 61 | 10
  Dengue Virus Serotype 4: 28 days Post-injection 2 | 89.6 [55.9 to 144] | 88.8 [56.0 to 141] | 223 [65.3 to 763]
  Dengue Virus Serotype 4: Pre-injection 3: number analyzed (Participants) | 51 | 60 | 9
  Dengue Virus Serotype 4: Pre-injection 3 | 40.0 [25.9 to 61.6] | 68.3 [45.0 to 104] | 146 [40.0 to 531]
  Dengue Virus Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 52 | 59 | 9
  Dengue Virus Serotype 4: 28 days Post-injection 3 | 51.7 [35.1 to 76.2] | 78.5 [54.3 to 114] | 182 [103 to 319]

8. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each Dengue Virus Serotype Following Each Injection With CYD Dengue Vaccine: Group 1, Group 2 and Group 3 (FV Non-Immune Participants)
Description: GMTs of antibodies against each dengue virus serotype (parental strain) was assessed using the dengue PRNT. FV non-immune participants were defined as participants with titer < 10 (1/dilution) for all serotypes with parental dengue virus strains (sera tested by PRNT) and with titer <10 (1/dilution) for YF virus (using sera with PRNT80 result).
Time Frame: Pre-injection 1, 2, 3 and 28 days post-injection 1, 2 and 3
Population: Analysis was performed on Full Analysis Set. Here, Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected, analyzed for Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3
Number analyzed (Participants) | 54 | 54 | 103
Titer (1/dilution)
  Dengue Virus Serotype 1: Pre-injection 1 | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0.
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 7.31 [5.79 to 9.23] | 8.18 [6.22 to 10.8] | 7.50 [6.30 to 8.92]
  Dengue Virus Serotype 1: Pre-injection 2: number analyzed (Participants) | 51 | 53 | 100
  Dengue Virus Serotype 1: Pre-injection 2 | 6.73 [5.49 to 8.23] | 10.1 [7.40 to 13.7] | 7.76 [6.46 to 9.32]
  Dengue Virus Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 48 | 53 | 90
  Dengue Virus Serotype 1: 28 days Post-injection 2 | 13.9 [9.64 to 20.2] | 13.0 [9.12 to 18.5] | 10.9 [8.55 to 14.0]
  Dengue Virus Serotype 1: Pre-injection 3: number analyzed (Participants) | 47 | 50 | 84
  Dengue Virus Serotype 1: Pre-injection 3 | 6.71 [5.54 to 8.13] | 8.97 [6.70 to 12.0] | 10.8 [8.52 to 13.8]
  Dengue Virus Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 42 | 49 | 84
  Dengue Virus Serotype 1: 28 days Post-injection 3 | 13.9 [9.49 to 20.4] | 14.4 [10.1 to 20.7] | 18.5 [13.9 to 24.8]
  Dengue Virus Serotype 2: Pre-injection 1 | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0.
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 18.5 [11.8 to 28.9] | 15.8 [10.4 to 23.9] | 10.3 [8.26 to 13.0]
  Dengue Virus Serotype 2: Pre-injection 2: number analyzed (Participants) | 50 | 53 | 100
  Dengue Virus Serotype 2: Pre-injection 2 | 18.9 [11.6 to 30.7] | 34.6 [20.4 to 58.6] | 11.6 [8.87 to 15.1]
  Dengue Virus Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 48 | 53 | 90
  Dengue Virus Serotype 2: 28 days Post-injection 2 | 47.8 [31.0 to 73.7] | 58.8 [36.5 to 94.8] | 30.8 [22.3 to 42.6]
  Dengue Virus Serotype 2: Pre-injection 3: number analyzed (Participants) | 47 | 51 | 86
  Dengue Virus Serotype 2: Pre-injection 3 | 18.2 [12.0 to 27.7] | 32.4 [21.5 to 48.9] | 23.1 [16.3 to 32.9]
  Dengue Virus Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 42 | 49 | 84
  Dengue Virus Serotype 2: 28 days Post-injection 3 | 42.1 [27.9 to 63.4] | 51.4 [32.8 to 80.6] | 46.4 [33.8 to 63.6]
  Dengue Virus Serotype 3: Pre-injection 1 | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0.
  Dengue Virus Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 54 | 52 | 103
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 22.2 [13.6 to 36.2] | 30.7 [18.8 to 49.9] | 8.00 [6.60 to 9.71]
  Dengue Virus Serotype 3: Pre-injection 2: number analyzed (Participants) | 51 | 53 | 100
  Dengue Virus Serotype 3: Pre-injection 2 | 13.5 [8.76 to 20.8] | 27.8 [17.3 to 44.8] | 9.06 [7.18 to 11.4]
  Dengue Virus Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 48 | 53 | 90
  Dengue Virus Serotype 3: 28 days Post-injection 2 | 30.3 [19.5 to 46.8] | 54.1 [33.3 to 87.8] | 18.5 [13.6 to 25.2]
  Dengue Virus Serotype 3: Pre-injection 3: number analyzed (Participants) | 47 | 50 | 86
  Dengue Virus Serotype 3: Pre-injection 3 | 19.8 [13.5 to 29.1] | 27.2 [18.3 to 40.3] | 17.5 [12.9 to 23.6]
  Dengue Virus Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 42 | 48 | 83
  Dengue Virus Serotype 3: 28 days Post-injection 3 | 46.9 [30.9 to 71.2] | 47.3 [32.5 to 69.0] | 30.2 [22.8 to 40.1]
  Dengue Virus Serotype 4: Pre-injection 1 | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0. | 5.00 [NA to NA] — The CI of Geometric Mean was not calculated when SD = 0.
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 54 | 52 | 102
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 197 [90.9 to 428] | 229 [107 to 488] | 20.5 [14.3 to 29.4]
  Dengue Virus Serotype 4: Pre-injection 2: number analyzed (Participants) | 50 | 52 | 100
  Dengue Virus Serotype 4: Pre-injection 2 | 54.4 [31.6 to 93.5] | 135 [67.5 to 268] | 18.2 [12.6 to 26.3]
  Dengue Virus Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 48 | 52 | 90
  Dengue Virus Serotype 4: 28 days Post-injection 2 | 122 [77.3 to 193] | 145 [83.0 to 253] | 42.8 [29.2 to 62.7]
  Dengue Virus Serotype 4: Pre-injection 3: number analyzed (Participants) | 47 | 49 | 85
  Dengue Virus Serotype 4: Pre-injection 3 | 62.8 [39.2 to 101] | 82.9 [48.2 to 143] | 47.8 [34.2 to 66.7]
  Dengue Virus Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 42 | 48 | 83
  Dengue Virus Serotype 4: 28 days Post-injection 3 | 91.8 [63.3 to 133] | 89.2 [53.3 to 149] | 71.2 [52.0 to 97.7]

9. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following Each Injection With CYD Dengue Vaccine: Group 1, Group 2 and Group 3 (FV Immune Participants)
Description: Seropositivity against each dengue virus serotypes (parental strains) was assessed using the dengue PRNT. Seropositive participants were defined as the participants with neutralizing antibody titer >=10 (1/dilution). FV immune participants at baseline were defined as participants with titer >= 10 (1/dilution) for at least 1 serotype with parental dengue virus strain (sera tested by PRNT) or with titer >=10 (1/dilution) for YF virus (sera with PRNT80 result).
Time Frame: Pre-injection 1, 2, 3 and 28 days post-injection 1, 2 and 3
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3
Number analyzed (Participants) | 63 | 65 | 11
percentage of participants
  Dengue Virus Serotype 1: Pre-injection 1 | 3.2 | 4.6 | 18.2
  Dengue Virus Serotype 1: 28 days Post-injection 1: number analyzed (Participants) | 63 | 64 | 11
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 47.6 | 26.6 | 45.5
  Dengue Virus Serotype 1: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 1: Pre-injection 2 | 51.8 | 38.5 | 54.5
  Dengue Virus Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 53 | 63 | 10
  Dengue Virus Serotype 1: 28 days Post-injection 2 | 67.9 | 61.9 | 70.0
  Dengue Virus Serotype 1: Pre-injection 3: number analyzed (Participants) | 51 | 58 | 9
  Dengue Virus Serotype 1: Pre-injection 3 | 45.1 | 36.2 | 55.6
  Dengue Virus Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 51 | 59 | 9
  Dengue Virus Serotype 1: 28 days Post-injection 3 | 54.9 | 61.0 | 88.9
  Dengue Virus Serotype 2: Pre-injection 1 | 1.6 | 4.6 | 27.3
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 79.4 | 69.2 | 81.8
  Dengue Virus Serotype 2: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 2: Pre-injection 2 | 75.0 | 75.4 | 72.7
  Dengue Virus Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 53 | 63 | 10
  Dengue Virus Serotype 2: 28 days Post-injection 2 | 88.7 | 95.2 | 100.0
  Dengue Virus Serotype 2: Pre-injection 3: number analyzed (Participants) | 51 | 60 | 9
  Dengue Virus Serotype 2: Pre-injection 3 | 70.6 | 86.7 | 88.9
  Dengue Virus Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 52 | 59 | 9
  Dengue Virus Serotype 2: 28 days Post-injection 3 | 84.6 | 94.9 | 100.0
  Dengue Virus Serotype 3: Pre-injection 1 | 4.8 | 7.7 | 54.5
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 74.6 | 66.2 | 100.0
  Dengue Virus Serotype 3: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 3: Pre-injection 2 | 80.4 | 70.8 | 81.8
  Dengue Virus Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 53 | 63 | 10
  Dengue Virus Serotype 3: 28 days Post-injection 2 | 90.6 | 92.1 | 100.0
  Dengue Virus Serotype 3: Pre-injection 3: number analyzed (Participants) | 51 | 60 | 9
  Dengue Virus Serotype 3: Pre-injection 3 | 74.5 | 85.0 | 77.8
  Dengue Virus Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 52 | 59 | 9
  Dengue Virus Serotype 3: 28 days Post-injection 3 | 84.6 | 94.9 | 88.9
  Dengue Virus Serotype 4: Pre-injection 1 | 12.7 | 1.5 | 36.4
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 61 | 65 | 11
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 65.6 | 61.5 | 90.9
  Dengue Virus Serotype 4: Pre-injection 2: number analyzed (Participants) | 56 | 65 | 11
  Dengue Virus Serotype 4: Pre-injection 2 | 76.8 | 63.1 | 90.9
  Dengue Virus Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 53 | 61 | 10
  Dengue Virus Serotype 4: 28 days Post-injection 2 | 81.1 | 78.7 | 100.0
  Dengue Virus Serotype 4: Pre-injection 3: number analyzed (Participants) | 51 | 60 | 9
  Dengue Virus Serotype 4: Pre-injection 3 | 74.5 | 76.7 | 88.9
  Dengue Virus Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 52 | 59 | 9
  Dengue Virus Serotype 4: 28 days Post-injection 3 | 82.7 | 88.1 | 100.0

10. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following Each Injection With CYD Dengue Vaccine: Group 1, Group 2 and Group 3 (FV Non-Immune Participants)
Description: Seropositivity against each dengue virus serotypes (parental strains) was assessed using the dengue PRNT. Seropositive participants were defined as the participants with neutralizing antibody titer >=10 (1/dilution). FV non-immune participants were defined as participants with titer < 10 (1/dilution) for all serotypes with parental dengue virus strains (sera tested by PRNT) and with titer <10 (1/dilution) for YF virus (using sera with PRNT80 result).
Time Frame: Pre injection 1, 2, 3 and 28 days post injection 1, 2 and 3
Population: Analysis was performed on Full Analysis Set. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Group 4.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3
Number analyzed (Participants) | 54 | 54 | 103
percentage of participants
  Dengue Virus Serotype 1: Pre-injection 1 | 0.0 | 0.0 | 0.0
  Dengue Virus Serotype 1: 28 days Post-injection 1 | 18.5 | 22.2 | 19.4
  Dengue Virus Serotype 1: Pre-injection 2: number analyzed (Participants) | 51 | 53 | 100
  Dengue Virus Serotype 1: Pre-injection 2 | 17.6 | 32.1 | 22.0
  Dengue Virus Serotype 1: 28 days Post-injection 2: number analyzed (Participants) | 48 | 53 | 90
  Dengue Virus Serotype 1: 28 days Post-injection 2 | 47.9 | 41.5 | 36.7
  Dengue Virus Serotype 1: Pre-injection 3: number analyzed (Participants) | 47 | 50 | 84
  Dengue Virus Serotype 1: Pre-injection 3 | 19.1 | 28.0 | 39.3
  Dengue Virus Serotype 1: 28 days Post-injection 3: number analyzed (Participants) | 42 | 49 | 84
  Dengue Virus Serotype 1: 28 days Post-injection 3 | 50.0 | 51.0 | 59.5
  Dengue Virus Serotype 2: Pre-injection 1 | 0.0 | 0.0 | 0.0
  Dengue Virus Serotype 2: 28 days Post-injection 1 | 48.1 | 40.7 | 33.0
  Dengue Virus Serotype 2: Pre-injection 2: number analyzed (Participants) | 50 | 53 | 100
  Dengue Virus Serotype 2: Pre-injection 2 | 46.0 | 60.4 | 33.0
  Dengue Virus Serotype 2: 28 days Post-injection 2: number analyzed (Participants) | 48 | 53 | 90
  Dengue Virus Serotype 2: 28 days Post-injection 2 | 83.3 | 79.2 | 68.9
  Dengue Virus Serotype 2: Pre-injection 3: number analyzed (Participants) | 47 | 51 | 86
  Dengue Virus Serotype 2: Pre-injection 3 | 55.3 | 72.5 | 57.0
  Dengue Virus Serotype 2: 28 days Post-injection 3: number analyzed (Participants) | 42 | 49 | 84
  Dengue Virus Serotype 2: 28 days Post-injection 3 | 83.3 | 79.6 | 83.3
  Dengue Virus Serotype 3: Pre-injection 1 | 0.0 | 0.0 | 0.0
  Dengue Virus Serotype 3: 28 days Post-injection 1: number analyzed (Participants) | 54 | 52 | 103
  Dengue Virus Serotype 3: 28 days Post-injection 1 | 50.0 | 61.5 | 21.4
  Dengue Virus Serotype 3: Pre-injection 2: number analyzed (Participants) | 51 | 53 | 100
  Dengue Virus Serotype 3: Pre-injection 2 | 41.2 | 60.4 | 26.0
  Dengue Virus Serotype 3: 28 days Post-injection 2: number analyzed (Participants) | 48 | 53 | 90
  Dengue Virus Serotype 3: 28 days Post-injection 2 | 68.8 | 75.5 | 52.2
  Dengue Virus Serotype 3: Pre-injection 3: number analyzed (Participants) | 47 | 50 | 86
  Dengue Virus Serotype 3: Pre-injection 3 | 63.8 | 68.0 | 50.0
  Dengue Virus Serotype 3: 28 days Post-injection 3: number analyzed (Participants) | 42 | 48 | 83
  Dengue Virus Serotype 3: 28 days Post-injection 3 | 85.7 | 85.4 | 73.5
  Dengue Virus Serotype 4: Pre-injection 1 | 0.0 | 0.0 | 0.0
  Dengue Virus Serotype 4: 28 days Post-injection 1: number analyzed (Participants) | 54 | 52 | 102
  Dengue Virus Serotype 4: 28 days Post-injection 1 | 70.4 | 75.0 | 46.1
  Dengue Virus Serotype 4: Pre-injection 2: number analyzed (Participants) | 50 | 52 | 100
  Dengue Virus Serotype 4: Pre-injection 2 | 66.0 | 73.1 | 41.0
  Dengue Virus Serotype 4: 28 days Post-injection 2: number analyzed (Participants) | 48 | 52 | 90
  Dengue Virus Serotype 4: 28 days Post-injection 2 | 87.5 | 82.7 | 67.8
  Dengue Virus Serotype 4: Pre-injection 3: number analyzed (Participants) | 47 | 49 | 85
  Dengue Virus Serotype 4: Pre-injection 3 | 80.9 | 79.6 | 77.6
  Dengue Virus Serotype 4: 28 days Post-injection 3: number analyzed (Participants) | 42 | 48 | 83
  Dengue Virus Serotype 4: 28 days Post-injection 3 | 95.2 | 83.3 | 84.3

11. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, Swelling) Following Any Vaccination With CYD Dengue Vaccine (Administered With or Without Yellow Fever Vaccine) or Yellow Fever Vaccine
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Grade 3 reactions: Pain: significant; prevents daily activity; Erythema and Swelling: >100 mm.
Time Frame: Within 7 days after any injection
Population: Analysis was performed on Safety Analysis set which included participants who received at least one injection of CYD dengue vaccine or YF vaccine. Here, "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- CYD Dengue Vaccine: Group 1: Participants received 3 doses of CYD dengue vaccine ; one each at 0, 6 and 12 months.
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3 | Yellow Fever Vaccine: Group 4
Number analyzed (Participants) | 118 | 119 | 115 | 27
Participants
  Any Injection site Pain: CYD Dengue Vaccine | 44 | 59 | 51 | NA — CYD Dengue vaccine was not administered to the specified group.
  Grade 3 Pain: CYD Dengue Vaccine | 0 | 3 | 1 | NA — CYD Dengue vaccine was not administered to the specified group.
  Any Injection site Pain: Yellow Fever Vaccine | NA — Yellow Fever vaccine was not administered to the specified group. | NA — Yellow Fever vaccine was not administered to the specified group. | 53 | 10
  Grade 3 Pain: Yellow Fever Vaccine | NA — Yellow Fever vaccine was not administered to the specified group. | NA — Yellow Fever vaccine was not administered to the specified group. | 1 | 0
  Any Injection site Erythema: CYD Dengue Vaccine | 5 | 10 | 1 | NA — CYD Dengue vaccine was not administered to the specified group.
  Grade 3 Erythema: CYD Dengue Vaccine | 0 | 0 | 0 | NA — CYD Dengue vaccine was not administered to the specified group.
  Any Injection site Erythema: Yellow Fever Vaccine | NA — Yellow Fever vaccine was not administered to the specified group. | NA — Yellow Fever vaccine was not administered to the specified group. | 5 | 0
  Grade 3 Erythema: Yellow Fever Vaccine | NA — Yellow Fever vaccine was not administered to the specified group. | NA — Yellow Fever vaccine was not administered to the specified group. | 0 | 0
  Any Injection site Swelling: CYD Dengue Vaccine | 5 | 2 | 0 | NA — CYD Dengue vaccine was not administered to the specified group.
  Grade 3 Swelling: CYD Dengue Vaccine | 0 | 0 | 0 | NA — CYD Dengue vaccine was not administered to the specified group.
  Any Injection site Swelling: Yellow Fever Vaccine | NA — Yellow Fever vaccine was not administered to the specified group. | NA — Yellow Fever vaccine was not administered to the specified group. | 2 | 0
  Grade 3 Swelling: Yellow Fever Vaccine | NA — Yellow Fever vaccine was not administered to the specified group. | NA — Yellow Fever vaccine was not administered to the specified group. | 0 | 0

12. Secondary Outcome: Number of Participants Reporting Solicited Systemic Reactions (Fever, Headache, Malaise, Myalgia, Asthenia) Following Any Vaccination With CYD Dengue Vaccine (Administered With or Without Yellow Fever Vaccine) or Yellow Fever Vaccine
Description: Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Grade 3 reactions: Fever: >= 39.0°C; Headache, Malaise, Myalgia, and Asthenia: significant; prevents daily activity.
Time Frame: Within 14 days after any injection
Population: Analysis was performed on Safety Analysis Set. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3 | Yellow Fever Vaccine: Group 4
Number analyzed (Participants) | 120 | 120 | 119 | 30
Participants
  Fever: Any Grade: number analyzed (Participants) | 117 | 119 | 115 | 26
  Fever: Any Grade | 7 | 5 | 4 | 1
  Fever: Grade 3: number analyzed (Participants) | 117 | 119 | 115 | 26
  Fever: Grade 3 | 1 | 1 | 0 | 0
  Headache: Any Grade: number analyzed (Participants) | 118 | 119 | 115 | 27
  Headache: Any Grade | 59 | 60 | 64 | 11
  Headache: Grade 3: number analyzed (Participants) | 118 | 119 | 115 | 27
  Headache: Grade 3 | 4 | 5 | 6 | 1
  Malaise: Any Grade: number analyzed (Participants) | 118 | 119 | 115 | 27
  Malaise: Any Grade | 63 | 53 | 53 | 12
  Malaise: Grade 3: number analyzed (Participants) | 118 | 119 | 115 | 27
  Malaise: Grade 3 | 10 | 8 | 10 | 3
  Myalgia: Any Grade: number analyzed (Participants) | 118 | 119 | 115 | 27
  Myalgia: Any Grade | 51 | 47 | 54 | 8
  Myalgia: Grade 3: number analyzed (Participants) | 118 | 119 | 115 | 27
  Myalgia: Grade 3 | 6 | 3 | 9 | 2
  Asthenia: Any Grade: number analyzed (Participants) | 118 | 119 | 115 | 27
  Asthenia: Any Grade | 41 | 36 | 40 | 9
  Asthenia: Grade 3: number analyzed (Participants) | 118 | 119 | 115 | 27
  Asthenia: Grade 3 | 6 | 5 | 6 | 2

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 28 days after each dose of CYD dengue vaccine and/or YF vaccine. Solicited Reaction (SR) data were collected within 7 and 14 days after each and any vaccination. Serious adverse event (SAE) data were collected throughout the study (up to 18 months after the first injection).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | CYD Dengue Vaccine: Group 1 | CYD Dengue Vaccine: Group 2 | CYD Dengue and Yellow Fever Vaccine: Group 3 | Yellow Fever Vaccine: Group 4
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/119 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/120 | 4/120 | 5/119 | 0/30
Other Adverse Events (participants affected / at risk) | 91/120 | 92/120 | 92/119 | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine: Group 1 (N=120) | CYD Dengue Vaccine: Group 2 (N=120) | CYD Dengue and Yellow Fever Vaccine: Group 3 (N=119) | Yellow Fever Vaccine: Group 4 (N=30)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blighted Ovum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine: Group 1 (N=120) | CYD Dengue Vaccine: Group 2 (N=120) | CYD Dengue and Yellow Fever Vaccine: Group 3 (N=119) | Yellow Fever Vaccine: Group 4 (N=30)
Nausea (Gastrointestinal disorders) | 4 (5) | 7 (7) | 1 (1) | 0 (0)
Asthenia (General disorders) | 41 (57) | 36 (61) | 40 (57) | 9 (9)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Injection Site Erythema (General disorders) | 5 (5) | 10 (11) | 5 (6) | 0 (0)
Injection Site Pain (General disorders) | 44 (71) | 59 (97) | 63 (138) | 10 (10)
Malaise (General disorders) | 63 (92) | 53 (93) | 53 (77) | 12 (12)
Pyrexia (General disorders) | 7 (7) | 6 (6) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) | 7 (8) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 51 (75) | 47 (78) | 54 (91) | 8 (8)
Headache (Nervous system disorders) | 60 (90) | 61 (110) | 64 (110) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 7 (7) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.